CLINICAL TRIAL: NCT00353847
Title: A Randomized, Single Blind, Controlled Clinical Trial to Evaluate the Pain Relief Efficacy, Functional Improvement and Safety of Acupuncture in Patients With Chronic Low Back Pain
Brief Title: Acupuncture for Treatment of Chronic LBP, RCT, Single Blinded
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYD-06
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2006-11-16 (Estimated); Status verified 2006-06

CONDITIONS: Chronic Low Back Pain
Keywords: acupuncture, RCTs, chronic LBP
MeSH Terms: interventions — Acupuncture Therapy

INTERVENTIONS:
Device: Acupuncture

SUMMARY:
The purpose of this study is to determine whether acupuncture is effective and safe in the treatment of chronic LBP.

DETAILED DESCRIPTION:
The purpose of this study is as follows:

1. pain : VAS
2. Function : Roland Disability Scale
3. Side effect
4. Validity

ELIGIBILITY:
Inclusion Criteria:

* Having chronic, non-specific, LBP of at least 3 months' duration over 20 years old.
* Back pain must be the chief complaint
* Having normal neurological test
* Having signature voluntarily an IRB-approved consent form at enrollment

Exclusion Criteria:

* Potential spinal disease (e.g. a spinal tumor, infection or fracture etc)
* Other diseases (e.g. bleeding disease, dementia,epilepsy, neurogenic disorder etc)
* Planned or got lumbar surgery
* The prior use of acupuncture within the past 6 months
* Inflammatory arthritis
* The current use of systematic corticosteroids, narcotics, anticoagulants, muscle relaxants
* The involvement in legal problem related to LBP
* Refusal to be randomized

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-07

PRIMARY OUTCOMES:
Visual Analogue Scale, RDQ scale

SECONDARY OUTCOMES:
Patient Global Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Youngdal Kwon, MD, Ph.D, Principal Investigator — Professor of College of Oriental Medicine, Wonkwang University
Locations (1):
- Wonkwang University Hospital, Gwangju, Gwangju, South Korea